CLINICAL TRIAL: NCT00258440
Title: A Pilot Trial of Extended Interval Dosing of Epoetin Alfa (Procrit®) for the Treatment of Anemia in Oncology Patients
Brief Title: Epoetin Alfa in Treating Patients With Anemia Who Are Undergoing Chemotherapy for Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor discontinued funding of the study
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Ortho Biotech, Inc. (Industry)
Responsible Party: Principal Investigator, Joseph Bubalo, PharmD, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000445450; OHSU-ONC-03017-LP (Other: OHSU Knight Cancer Institute); OHSU-1616 (Other: OHSU IRB); OHSU-7754 (Other: OHSU Knight Cancer Institute); ORTHO-ONC-03017-LP (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2005-11-23; First posted 2005-11-24 (Estimated); Results first posted 2011-05-26 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Anemia; Fatigue; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: fatigue; anemia; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Anemia; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Weekly Procrit (epoetin alfa) dosing (Active Comparator): Weekly dosing schedule subjects will get the study drug once every week until the end of the study.
  Interventions: Drug: Weekly procrit dosing
- Interval Dosing (epoetin alfa) PK Group (Experimental): Interval-dosing schedule subjects will get the study drug once every week until hematocrit is greater than 36% or Hemoglobin reaches a value of 12 g/dl, then they will get study drug once every other week. Subjects who consented to pharmacokinetic testing
  Interventions: Drug: Interval Dosing
- Interval Dosing (epoetin alfa) Non PK Group (Experimental): Interval-dosing schedule subjects will get the study drug once every week until hematocrit is greater than 36% or Hemoglobin reaches a value of 12 g/dl, then they will get study drug once every other week. Subjects who did not consent to pharmacokinetic testing.
  Interventions: Drug: Interval Dosing

INTERVENTIONS:
Drug: Weekly procrit dosing — The dose is standard of care, the investigational piece is the dosing schedule itself. Either weekly or Interval-dosing schedule subjects will get the study drug once every week until hematocrit is greater than 36% or Hemoglobin reaches a value of 12 g/dl, then they will get study drug once every other week.
  Arms: Weekly Procrit (epoetin alfa) dosing
Drug: Interval Dosing — The dosing of Procrit is standard of care, it is the schedule that is the investigational piece.
  Arms: Interval Dosing (epoetin alfa) Non PK Group; Interval Dosing (epoetin alfa) PK Group

SUMMARY:
RATIONALE: Epoetin alfa may cause the body to make more red blood cells. It is used to treat anemia caused by cancer and chemotherapy. It may also help relieve fatigue in patients with anemia.

PURPOSE: This randomized clinical trial is studying how well epoetin alfa works in treating patients with anemia who are undergoing chemotherapy for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy, in terms of maintenance of target hemoglobin and hematocrit levels, of interval dosing with epoetin alfa in treating patients with anemia undergoing chemotherapy for nonhematologic cancer.

Secondary

* Determine the pharmacokinetics and pharmacodynamics of this drug in these patients.
* Correlate hemoglobin and hematocrit response with patient age (> 65 years vs < 65 years) in patients treated with this drug.
* Determine quality of life of patients treated with this drug.
* Determine the adverse effects of this drug in these patients.
* Determine the change over time of symptom and quality of life variables (e.g., fatigue) in patients treated with this drug.

OUTLINE: This is a partially randomized, pilot study. Patients are stratified according to age (< 65 years vs ≥ 65 years). Patients are assigned to 1 of 2 treatment groups based on participation in the pharmacokinetic (PK) portion of the study.

* Group 1 (PK study, initial therapy): Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Five patients receive epoetin alfa subcutaneously (SC) once weekly. Treatment continues for 24 weeks in the absence of unacceptable toxicity.
  * Arm II: Five patients receive epoetin alfa SC once weekly until hematocrit is > 36% OR hemoglobin reaches a value of 12 g/dL. Patients then proceed to maintenance therapy.

Patients in both arms also undergo PK sampling periodically during study treatment.

* Group 2 (non-PK study, initial therapy): Fifteen patients receive epoetin alfa SC once weekly until hematocrit is > 36% OR hemoglobin reaches a value of 12 g/dL. Patients then proceed to maintenance therapy.
* Maintenance therapy: Patients receive epoetin alfa SC once every other week for up to 24 weeks of total treatment (including both initial therapy and maintenance therapy). Patients whose blood counts fall below the critical levels are placed on a weekly dosing schedule. Patients whose blood counts rise too high discontinue study drug until blood counts are reduced.

Quality of life (including fatigue) is assessed at baseline and then every 4 weeks for 28 weeks.

After completion of study therapy, patients are followed at 4 weeks.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study.

ELIGIBILITY:
ELIGIBILITY CRITERIA

* 18 years of age or greater
* Must have Hb less than 11 g/dl and normal hematopoesis
* Must have non-myeloid malignancies treated with myelosuppressive therapy *Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Must have a life expectancy of 6 months or greater
* Must have adequate liver function (bilirubin less than or equal to 2.0 mg) and renal function (creatinine less than or equal to 2.0 mg)
* Must have normal serum folate and vitamin B12 levels or be receiving replacement therapy
* Must be iron replete (transferring saturation great than or equal to 20 percent and ferritin greater than or equal to 100 mg/ml) or be receiving replacement therapy
* Must be able to fully comprehend and give written consent.
* Female patients with reproductive potential must be practicing an effective method of birth control (e.g., abstinence, prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, surgical sterilization) before entry and throughout the study.
* Female patients with reproductive potential must have a negative serum human chorionic gonadotropin (HCG) pregnancy test at screening (within 7 days before the first dose of study drug)

Exclusion criteria

* Patient has uncontrolled hypertension
* Patient has history of symptomatic cardiac disease
* Patient has serious intercurrent illness
* The patient is pregnant, has a positive serum HCG or is lactating Patient has known hypersensitivity to mammalian cell-derived products or human albumin.
* Patient has diagnosis of polycythemia vera, chronic myelogenous leukemia, myelodysplastic syndrome
* May not be due for transplant within 24 weeks
* Anemia due to factors other than cancer.
* History of a thrombotic vascular event.
* History of seizures
* Patient has received a red blood cell growth factor (epoetin alfa or darbepoetin) within the last 60 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2003-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Bubalo, PharmD, BCPS, BCOP, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were adults age >=18yrs, with solid tumors, and who received treatment. A total of 25 subjects were recruited. Potential study subjects were seen in a routine clinical setting or referred for study purposes. The PI, physician or the research nurse approached subject and to get informed consent, as well as screen for eligibility.
Groups:
- Weekly Procrit (Epoetin Alfa) Dosing: Patients receive epoetin alfa subcutaneously (SC) once weekly. Treatment continues for 24 weeks in the absence of unacceptable toxicity. Patients then proceed to maintenance therapy.
- Interval Dosing (Epoetin Alfa) PK Group: Patients receive epoetin alfa SC once weekly until hematocrit is > 36% OR hemoglobin reaches a value of 12 g/dL. Patients then proceed to maintenance therapy. Patients who have consented to pharmacokinetics (PK) testing.
- Interval Dosing (Epoetin Alfa) Non PK Group: Patients receive epoetin alfa SC once weekly until hematocrit is > 36% OR hemoglobin reaches a value of 12 g/dL. Patients then proceed to maintenance therapy. Patients who have NOT consented to pharmacokinetics (PK) testing.
Period: Overall Study
Arm/Group | Weekly Procrit (Epoetin Alfa) Dosing | Interval Dosing (Epoetin Alfa) PK Group | Interval Dosing (Epoetin Alfa) Non PK Group
Started | 1 | 0 | 6
Completed | 1 | 0 | 5
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Weekly Procrit (Epoetin Alfa) Dosing | Interval Dosing (Epoetin Alfa) PK Group | Interval Dosing (Epoetin Alfa) Non PK Group | Total
Number analyzed (Participants) | 1 | 0 | 6 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0 | 0
  Between 18 and 65 years | 1 |  | 6 | 7
  >=65 years | 0 |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 5 | 5
  Male | 1 |  | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 6 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects That Maintained Target Hemoglobin Level (11-12 g/dL) Maintenance Weekly for 12 Weeks
Time Frame: 12 weeks
Population: Due to low accrual numbers and the discontinuation of the study early a full analysis was not completed.
Measure: Number; unit: participants
Arm/Group | Weekly Procrit (Epoetin Alfa) Dosing | Interval Dosing (Epoetin Alfa) PK Group | Interval Dosing (Epoetin Alfa) Non PK Group
Number analyzed (Participants) | 1 | 0 | 6
participants | 0 [1 to 6] |  | 5

2. Secondary Outcome: Pharmacokinetics (PK) and Pharmacodynamics Assays That Measure Concentration of Erythropoietin in Serum.
Time Frame: every other week
Reporting Status: Not Posted

3. Secondary Outcome: Quality of Life at Baseline and Weeks 4, 8, 16, 24, and 28
Time Frame: weeks 4,8,16,24 and 28
Reporting Status: Not Posted

4. Secondary Outcome: Number of Adverse Events (AEs) Experienced as Measure of Safety and Tolerability.
Time Frame: On study, averaging 3 to 6 months.
Measure: Number; unit: events
Arm/Group | Weekly Procrit (Epoetin Alfa) Dosing | Interval Dosing (Epoetin Alfa) PK Group | Interval Dosing (Epoetin Alfa) Non PK Group
Number analyzed (Participants) | 1 | 0 | 6
events | 38 |  | 130

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for as long as the patient was on study. in some cases that was up to 6 months or as little as 3 months.
Arm/Group | Weekly Procrit (Epoetin Alfa) Dosing | Interval Dosing (Epoetin Alfa) PK Group | Interval Dosing (Epoetin Alfa) Non PK Group
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 1/6
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weekly Procrit (Epoetin Alfa) Dosing (N=1) | Interval Dosing (Epoetin Alfa) PK Group (N=0) | Interval Dosing (Epoetin Alfa) Non PK Group (N=6)
Failure to thrive, GI bleed, Malignant Hypercalcemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — Patient went on to comfort care due to tumor progression.
Fever Neutropenia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Subject experienced neutropenic fever and was admitted.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weekly Procrit (Epoetin Alfa) Dosing (N=1) | Interval Dosing (Epoetin Alfa) PK Group (N=0) | Interval Dosing (Epoetin Alfa) Non PK Group (N=6)
lymphopenia (Blood and lymphatic system disorders) | 1 (6) | 0 (0) | 5 (22)
Platelets (Blood and lymphatic system disorders) | 1 (6) | 0 (0) | 5 (21)
Leukocytes (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 2 (7)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (4) | 0 (0) | 5 (7)
Fatigue (General disorders) | 1 (2) | 0 (0) | 5 (8)
Nausea (General disorders) | 1 (1) | 0 (0) | 3 (8)
Abdominal bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal cramping (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Increasing abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pain upper abdomen (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain/tumor pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage, nose (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage, urine trace (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bilateral lower extremity edema (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thigh swelling (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Abnormal metabolic labs (Metabolism and nutrition disorders) | 1 (12) | 0 (0) | 5 (31)

LIMITATIONS AND CAVEATS:
Due to low accruals the sponsor decided to discontinue the study early. A full analysis was not completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No